CLINICAL TRIAL: NCT04792242
Title: Comparison Between Goal Directed Therapy and PCO2 Gap Algorithm Application on Outcome of High Risk Surgical Patients Undergoing Major Abdominal Surgeries
Brief Title: Effect of PCO2 Gap Algorithm Application on Outcome of High Risk Surgical Patients Undergoing Major Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Hassan Abdelsapour Abdelrazek, PhD Candidat, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SVU.MED.AIP029.4.1
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Major Abdominal Surgeries
MeSH Terms: interventions — Urinary Catheterization; Vascular Access Devices

STUDY DESIGN:
Intervention Model Description: case control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- goal directed therapy (Active Comparator): svo2,haematocrite value,urine output,mean arterial pressure and central venous pressure
  Interventions: Device: cv line insertion; Device: Urinary catheter insertion
- PCO2 gap algorithm (Active Comparator): PCO2 gap,haematocrite value,Spo2,cardiac index
  Interventions: Device: cv line insertion; Device: Urinary catheter insertion; Device: Arterial line

INTERVENTIONS:
Device: cv line insertion — Svo2 and central venous pressure measurements
Device: Urinary catheter insertion — urine output measurement
Device: Arterial line — Arterial blood gases measurment
  Arms: PCO2 gap algorithm

SUMMARY:
1. Primary (main):

   Comparison between goal directed therapy and PCO2 gap algorithm (carbon dioxide partial pressure venous arterial gap algorithm) application on 30 days mortality and organ dysfunction post operative
2. Secondary (subsidiary):

Comparison between goal directed therapy and PCO2 gap algorithm application on number of ventilator dependant days, number of days on vasopressors or inotropes length of ICU stay, length of hospital stay,

DETAILED DESCRIPTION:
High risk surgical participants in South valley university hospitals (teaching hospitals) who will undergo major abdominal surgeries will be included in research after giving written informed consent from the participants or from the patient's legal representative. The use of obtained data will be approved by local ethics committee.

All participants will be evaluated pre operatively and pre medicated according to protocols in our hospital, base line sequential organ failure (SOFA) score will be taken. General anesthesia for all patients will be carried on according to our local standards. As part of our routine hemodynamic monitoring during major surgery, all patients will be monitored with central venous (standard three-lumen catheter) and arterial catheters placed before the beginning of surgery. The central venous line will be positioned with the tip within the superior vena cava, and correct positioning will be verified by chest radiograph.

the participants will be divided randomly onto to groups using numerical system group A PCO2 gap algorithm(carbon dioxide partial pressure venous arterial gap) will be applied intraoperative and 12 h postoperative end point PCO2 gap 2-6mm Hg(appendix 1).

Group B goal directed therapy protocol which will include targets mean arterial blood pressure ( MAP) > 65 mmHg, central venous pressure(CVP) between 8-12 cmH2O , Haematocrite value more than 30, mixed venous oxygen saturation (Svo2) >75% and urine output more than >0.5 ml/kg/hr and will be applied intraoperative and 12 postoperative end point base deficit +/- 2(appendix 2 ).

All participants will be admitted to the ICU (intensive care unit) immediately after surgery .Standard postoperative monitoring will include: electrocardiograph (heart rate), invasive mean arterial pressure, pulse oxygen saturation and urine output then will be all managed according to their allocated group for 12 hours.

Outcomes in both groups will be recorded which will be number of ventilator dependant days, number of days on vasopressors or inotropes length of ICU stay, length of hospital stay, 30 days organ dysfunction, assessed by using the Sequential Organ Failure Assessment (SOFA) and 30 days mortality .

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for high-risk surgical patients used by Shoemaker and colleagues and adapted by Boyd and colleagues

Exclusion Criteria:

* patients who will refuse to continue on research patients who will not be admitted post operative in the ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Post operative mortality | 30 days
  early post operative mortality

SECONDARY OUTCOMES:
post operative organ failure | 30 days
  cardiac,renal,respiratory,renal central nervous system(CNS) failure by sequential organ failure(SOFA) score

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Luxor, Qena Governorate, Egypt